CLINICAL TRIAL: NCT05300828
Title: An Observational Study to Evaluate the Safety of the Combination Therapy of Genexol PM and Carboplatin as First-line Therapy for Ovarian Cancer Patients
Brief Title: Safety of Genexol PM and Carboplatin as First-line Therapy in Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Principal Investigator, Hee Seung Kim, Professor, Seoul National University Hospital
Other Study IDs: GENEXOL PM
Record Dates: First submitted 2022-03-19; First posted 2022-03-29 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Genexol PM: Genexol PM/carboplatin combination treatment is performed as an adjuvant treatment after cytoreductive surgery for newly diagnosed ovarian cancer.
  Interventions: Drug: Genexl PM

INTERVENTIONS:
Drug: Genexl PM — Every three weeks, after intravenous infusion of 260 mg/m2 for 3 hours, followed by carboplatin AUC 5 for 3 hours.

SUMMARY:
To evaluate the safety profile of Genexol PM combination with carboplatin for patients with newly diagnosed ovarian cancer. We hypothesized Genexol PM can be safely administered to newly diagnosed ovarian cancer patients compared to conventional paclitaxel/carboplatin combination therapy. Therefore, we will compare the prospective cohort with a historical comparison with patients administered paclitaxel/carboplatin and paclitaxel/carboplatin/bevacizumab combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Patients consented to participate
* Pathologically diagnosed ovarian cancer FIGO stage IC-IVB
* ECOG 0-2
* Patients with an expected survival of 3 months or more

Exclusion Criteria:

* History of paclitaxel or carboplatin hypersensitivity
* Inadequate bone marrow function (Neutrophil<1500/mm3, Platelet <100,000/mm3)
* Pregnancy or breast-feeding state
* Metachronous or synchronous malignancy
* Galactose intolerance, Lapp Lactase deficiency, or glucose-galactose malabsorption patients with genetic problems
* Other patients who were judged difficult to be included in this investigation by the investigator in charge

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients at tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2015-10-19 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants showing adverse events | From the time of treatment start date through 30 days following cessation of treatment
  Number of any adverse event assessed based on CTCAE 4.0

SECONDARY OUTCOMES:
Neurotoxicity | From the time of treatment start date through 30 days following cessation of treatment
  Number of participants showing grade 3/4 neurotoxicity assessed based on CTCAE 4.0
other toxicity | From the time of treatment start date through 30 days following cessation of treatment
  Number of participants showing grade 3/4 any toxicity assessed based on CTCAE 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Hee Seung Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Division of Gynecologic Oncology, Department of Obstetrics and Gynecology, Ajou University School of Medicine, Suwon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee SW, Kim YM, Cho CH, Kim YT, Kim SM, Hur SY, Kim JH, Kim BG, Kim SC, Ryu HS, Kang SB. An Open-Label, Randomized, Parallel, Phase II Trial to Evaluate the Efficacy and Safety of a Cremophor-Free Polymeric Micelle Formulation of Paclitaxel as First-Line Treatment for Ovarian Cancer: A Korean Gynecologic Oncology Group Study (KGOG-3021). Cancer Res Treat. 2018 Jan;50(1):195-203. doi: 10.4143/crt.2016.376. Epub 2017 Mar 21. PMID 28324920
- [Background] Lee SW, Kim YM, Kim YT, Kang SB. An open-label, multicenter, phase I trial of a cremophor-free, polymeric micelle formulation of paclitaxel combined with carboplatin as a first-line treatment for advanced ovarian cancer: a Korean Gynecologic Oncology Group study (KGOG-3016). J Gynecol Oncol. 2017 May;28(3):e26. doi: 10.3802/jgo.2017.28.e26. Epub 2016 Dec 19. PMID 28028994